## Title: Optimizing an mHealth Intervention to Change Food Purchasing Behaviors for Cancer Prevention NCT04947150

Document date: 3/25/21

## **Statistical Analyses**

We will run repeated measures ANOVAs that examined whether outcomes change across time (i.e., from baseline to post-treatment). Models also include the interaction effects of each intervention component (location triggered messaging, benefits of change, coach monitoring, and household support) and time to determine whether these components could enhance change. Each condition variable is coded as 0=OFF or 1=ON, and all conditions are included in a single model for each outcome. We also report and interpret effect sizes (partial eta squared;  $\eta^2$ ) in addition to p-values. Effect sizes are interpreted as meaningful if they are .06 or higher, indicating a medium effect. Post-hoc pairwise comparisons examine change in each guideline across time separately for each condition.